CLINICAL TRIAL: NCT06119880
Title: The Effect of PERT on Postoperative Complications and Physiological Status in Patients Undergoing Pancreaticoduodenectomy
Brief Title: The Effect of PERT on Patients Undergoing Pancreaticoduodenectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Weishen WANG, Principal Investigator, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HBP-RCT-004
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Exocrine Insufficiency; Pancreatic Enzyme Replacement Therapy; Pancreaticoduodenectomy
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PERT Group (Experimental): After surgery, resume diet and begin receiving standard PERT treatment (2 capsules per meal, 1 capsule per snack, taken with meals, starting at a dose of 40000 to 50000 units of lipase) for 8 weeks.
  Interventions: Drug: Pancreatin Enteric-coated Capsules
- Placebo Group (Placebo Comparator): Follow the routine treatment plan for pancreatic tumors during the perioperative period.
  Interventions: Other: Routine treatment plan

INTERVENTIONS:
Drug: Pancreatin Enteric-coated Capsules — pancreatic enzyme replacement therapy
  Arms: PERT Group
Other: Routine treatment plan — Routine treatment plan without PERT
  Arms: Placebo Group

SUMMARY:
A comprehensive perioperative nutrition management plan for pancreaticoduodenectomy, primarily based on pancreatic enzyme replacement therapy (PERT). A prospective randomized controlled study was conducted to comprehensively analyze the perioperative nutritional status of patients undergoing pancreaticoduodenectomy, with the aim of exploring:

1. The effect of PERT on postoperative complications and physiological status after pancreaticoduodenectomy;
2. The efficacy of PERT treatment on clinical symptoms, nutritional indicators, and quality of life (QOL) related to pancreatic exocrine dysfunction (PEI) after pancreaticoduodenectomy;
3. The personalized full process nutrition management strategies based on risk factor stratification.

ELIGIBILITY:
Inclusion Criteria:

* Gender unlimited, 18-80 years old;
* Patients undergoing pancreaticoduodenectomy due to various benign or malignant diseases;
* Voluntary testing with informed consent.

Exclusion Criteria:

* Pregnant women and lactating women
* Patients with distant metastasis based on tumor staging before surgery;
* Tumor recurrence;
* Refuse to sign the consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Abdominal Skeletal Muscle Index (SMI) | 8 weeks post-operation
  Measurement of abdominal skeletal muscle area at the third lumbar spine plane using abdominal plain scan CT and comparison of baseline level SMI change rate.

SECONDARY OUTCOMES:
Postoperative complications | 8 weeks post-operation
  postoperative pancreatic fistula, delayed gastric emptying, postoperative hypoproteinemia;
Nutritional indicators | 8 weeks post-operation
  Patient generated subjective global assessment (PG-SGA);

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China